CLINICAL TRIAL: NCT05678946
Title: The Effects of Integrated Face-to-face Rehabilitation and Telerehabilitation on the Well-being of Family Caregivers
Status: Completed | Type: Observational
Sponsor: Social Insurance Institution, Finland (Other)
Responsible Party: Sponsor
Other Study IDs: SocialII
Record Dates: First submitted 2012-06-07; First posted 2023-01-10 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Caregivers; Family Caregivers; Informal Caregivers
Keywords: rehabilitation; effects; effectiveness; telerehabilitation; family caregivers; informal caregivers; family caregivers burden
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Integrated face-to-face rehabilitation and telerehabilitation: Participation in integrated face-to-face rehabilitation and telerehabilitation services for family caregivers organized by the Social Insurance Institution of Finland (Kela)
  Interventions: Other: Integrated face-to-face rehabilitation and telerehabilitation
- Social Holidays: Participation in face-to-face Social Holidays for family caregivers organized by Maaseudun Terveys- ja Lomahuolto (MTLH), a non-profit organization
  Interventions: Other: Social Holidays
- Face-to-face rehabilitation: Participation in face-to-face rehabilitation services for family caregivers and the care recipients organized by Kela
  Interventions: Other: Face-to-face rehabilitation

INTERVENTIONS:
Other: Integrated face-to-face rehabilitation and telerehabilitation — Kela´s integrated face-to-face rehabilitation and telerehabilitation services for family caregivers include two 5-day periods of face-to-face rehabilitation and a 12-week telerehabilitation period between them. It is for those over the age of 18 who work as family caregivers on a daily basis and need support, tools, and coaching to understand and overcome the challenges posed by the care situation. Individual goals based on the GAS method are set, evaluated, and adjusted during the rehabilitation. The service, provided free of charge, is carried out in a Finnish rehabilitation centre and online over a period of 8 months, and it is implemented by a multidisciplinary team of rehabilitation experts. During the 12-week telerehabilitation period, the service providers utilise The Own Path, an acceptance and commitment therapy -based guided web intervention found beneficial for older Finnish family caregivers (Lappalainen et al. 2021). Telerehabilitation is independent of time and place.
  Groups: Integrated face-to-face rehabilitation and telerehabilitation
Other: Social Holidays — MTLH's Social Holidays for family caregivers are 5-day holidays in a Finnish hotel, spa, sports institute, or rehabilitation centre. The theme, content, and level of available assistance in Social Holidays vary, and the rehabilitation concept is lighter than that of Kela's rehabilitation services. Social Holidays include full-board accommodation and holiday activities, e.g. lectures, group discussions, instructed exercise, and a pampering treatment. MTLH organises Social Holidays for family caregivers as well as family caregivers and care recipients. The participants cover their travel expenses and pay a fixed sum of €125. Other than that, Social Holidays are provided free of charge. Social Holidays are intended for family caregivers who need recreational activities, rest, and peer support.
  Groups: Social Holidays
Other: Face-to-face rehabilitation — Kela's rehabilitation services for family caregivers and the care recipients include three 5-day periods of face-to-face rehabilitation, which are carried out in a Finnish rehabilitation centre over a 10-month period and implemented by a multidisciplinary team of rehabilitation experts. The rehabilitation services for family caregivers and the care recipients are provided free of charge. The service is intended for persons over the age of 18 who work as family caregivers on a daily basis with or without family caregiver support and who need support, tools, and coaching to understand and overcome the challenges posed by the care situation. Individual goals based on the GAS method are set, evaluated, and adjusted during the rehabilitation.
  Groups: Face-to-face rehabilitation

SUMMARY:
This controlled, non-randomized study (n=180) explores how participating in rehabilitation services for family caregivers affects the caregivers' mood, perceived quality of life, perceived burden of family care, and overall health. Rehabilitation services for family caregivers funded by the Social Insurance Institution of Finland (Kela) include two 5-day periods of face-to-face rehabilitation and a 12-week telerehabilitation period, which is based on The Own Path internet intervention and takes place between the face-to-face rehabilitation periods. The observed changes are compared to participating in two other services: 1) Social Holidays for family caregivers and 2) Kela's rehabilitation services for family caregivers and the family members they are caring for (care recipients).

ELIGIBILITY:
Inclusion Criteria:

* family caregiver
* being 18 years of age or older
* providing daily care for an adult family member
* participating in one of following:

  1. the Kela's integrated face-to-face rehabilitation and telerehabilitation service for family caregivers,
  2. the MTLH's face-to-face Social Holidays for family caregivers or
  3. the Kela's face-to-face rehabilitation services for family caregivers and care recipients
* willingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those starting in one of the following services during April 2022 and January 2023:
  1. the Kela's integrated face-to-face rehabilitation and telerehabilitation service for family caregivers,
  2. the MTLH's face-to-face Social Holidays for family caregivers or
  3. the Kela's face-to-face rehabilitation services for family caregivers and care recipients
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mood at 5 months and 8 months | Baseline (pre-intervention), 5 months (after the intervention), 8 months (3-month follow-up)
  assessed with the Beck's Depression Inventory (BDI-21)

SECONDARY OUTCOMES:
Change from baseline in Quality of life (QoL) at 5 months and 8 months | Baseline (pre-intervention), 5 months (after the intervention), 8 months (3-month follow-up)
  assessed with the World Health Organization Quality of Life Instrument (WHOQOL-BREF)
Change from baseline in perceived burden of family care (I) at 5 months and 8 months | Baseline (pre-intervention), 5 months (after the intervention), 8 months (3-month follow-up)
  assessed with the Carers of Older People in Europe (COPE) index
Change from baseline in perceived burden of family care (II) at 5 months and 8 months | Baseline (pre-intervention), 5 months (after the intervention), 8 months (3-month follow-up)
  assessed with the Adult Social Care Outcomes Toolkit (ASCOT) questionnaire
Change from baseline in overall health at 5 months and 8 months | Baseline (pre-intervention), 5 months (after the intervention), 8 months (3-month follow-up)
  assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) survey
Individual goal achievement | 5 months (after the intervention)
  assessed with the Goal Attainment Scaling method (GAS)

CONTACTS AND LOCATIONS:
Overall Officials: Saija Karinkanta, PhD, Principal Investigator — The Social Insurance Institution of Finland (Kela)
Locations (1):
- The Social Insurance Institution of Finlad, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lappalainen P, Pakkala I, Lappalainen R, Nikander R. Supported Web-Based Acceptance and Commitment Therapy for Older Family Caregivers (CareACT) Compared to Usual Care. Clin Gerontol. 2022 Jul-Sep;45(4):939-955. doi: 10.1080/07317115.2021.1912239. Epub 2021 Apr 15. PMID 33856279